CLINICAL TRIAL: NCT06660797
Title: Effect of Different Irrigation Activating Techniques on Irrigant Penetration Depth and Microbial Reduction in Root Canals (Clinical Study)
Brief Title: Irrigation Activating Techniques on Irrigant Penetration Depth and Microbial Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Samy Abd Elsabour Alfky, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Irrigation Activation
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Irrigation Activation; Endodontic Disease
Keywords: Different Irrigation Activating Techniques; primary Endodontic Infection cases
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group 1: Manual dynamic agitation by matching gutta-percha master cones (Active Comparator): matching gutta-percha master cones will be used in up and down motion 2mm amplitude at a frequency of 100 strokes during approximately 1 min in each prepared canal.
  Interventions: Other: Group1: A matching gutta-percha master cones will be used in up and down motion 2mm amplitude at a frequency of 100 strokes during approximately 1 min in each prepared canal.
- Group 3: Easy Clean system activation (Active Comparator): EC instrument coupled to the countrangle handpiece and operated with a micromotor at approximately 20,000 rotations per minute in continuous rotation.
  Interventions: Other: Group 3:EasyClean system activation : EC instrument coupled to the countrangle handpiece and operated with a micromotor at approximately 20,000 rotations per minute in continuous rotation.
- Group 2: XP-endo Finisher activation (Active Comparator): XP-endo Finisher used in continuous rotation for 1 minute accompanied with in-and-out movements of approximately 7-mm amplitude will be applied to the instrument according to the manufacturer's recommendations⁸
  Interventions: Other: Group2: XP-endo Finisher activation: The XP-endo Finisher instrument will be used in continuous rotation for 1 mintute

INTERVENTIONS:
Other: Group1: A matching gutta-percha master cones will be used in up and down motion 2mm amplitude at a frequency of 100 strokes during approximately 1 min in each prepared canal. — The first microbial sample (S1) will be taken from the root canal immediately after access cavity preparation and before chemomechanical preparation.Samples will be subjected to bacterial viable count using blood agar. After complete chemomechanical preparation, a second microbial samble (S2) will be taken and managed the same way as S1.After irrigation activation protocol by matching gutta percha master cone , S3 will be collected from each root canal and managed as S1, S2 to evaluate effect of activation techniques on microbial reduction ,canals will be dried with a matching paper point then 1 mL of Iohexol (omnipaque) contrast media will be injected 2mL shorter than WL and activated by a matching gutta percha master cone , a digital radiographic image will be obtained for each tooth with the same angulation as that for WL and then the distance between WL and maximum irrigant penetration will be measured and recorded using SIDEXIS-XG software.
  Arms: • Group 1: Manual dynamic agitation by matching gutta-percha master cones
Other: Group2: XP-endo Finisher activation: The XP-endo Finisher instrument will be used in continuous rotation for 1 mintute — The first microbial sample (S1) will be taken from the root canal immediately after access cavity preparation and before chemomechanical preparation.Samples will be subjected to bacterial viable count using blood agar. After complete chemomechanical preparation, a second microbial samble (S2) will be taken and managed the same way as S1.After irrigation activation protocol by XP-endo Finisher used in continuous rotation for 1 minute , S3 will be collected from each root canal and managed as S1, S2 to evaluate effect of activation techniques on microbial reduction ,canals will be dried with a matching paper point then 1 mL of Iohexol (omnipaque) contrast media will be injected 2mL shorter than WL and activated by a matching gutta percha master cone , a digital radiographic image will be obtained for each tooth with the same angulation as that for WL and then the distance between WL and maximum irrigant penetration will be measured and recorded using SIDEXIS-XG software.
  Arms: Group 2: XP-endo Finisher activation
Other: Group 3:EasyClean system activation : EC instrument coupled to the countrangle handpiece and operated with a micromotor at approximately 20,000 rotations per minute in continuous rotation. — after access cavity preparation and before chemomechanical preparation.Samples will be subjected to bacterial viable count using blood agar. After complete chemomechanical preparation, a second microbial samble (S2) will be taken and managed the same way as S1.After irrigation activation protocol by EasyClean system activation , S3 will be collected from each root canal and managed as S1, S2 to evaluate effect of activation techniques on microbial reduction ,canals will be dried with a matching paper point then 1 mL of Iohexol (omnipaque) contrast media will be injected 2mL shorter than WL and activated by a matching gutta percha master cone , a digital radiographic image will be obtained for each tooth with the same angulation as that for WL and then the distance between WL and maximum irrigant penetration will be measured and recorded using SIDEXIS-XG software.
  Arms: Group 3: Easy Clean system activation

SUMMARY:
This in-vivo study aim to evaluate effect of different irrigation activating techniques on Irrigant Penetration Depth and Microbial Reduction in root Canals

DETAILED DESCRIPTION:
Chemomechanical preparation with removal of infected tissues and microbial biofilms is the corner stone of root canal treatment. Since mechanical instrumentation alone cannot adequately disinfect root canals, complete cleaning and shaping involves irrigation with chemicals together with mechanical instrumentation.

In addition to shaping the root canal, the aim of chemical-mechanical preparation of root canals is to eliminate vital or necrotic tissue, microorganisms and their products, and dentin debris that result from instrumentation. However, the complexity of root canal anatomy together with microbial infection hinder this purpose.

Primary endodontic infection is characterized by the presence of a wide range of microbial diversity dominated by anaerobes. The polymicrobial profile of pulp infection involves both Gram-positive and Gram-negative bacterial species.

Besides, the apical third of the root canal system typically has a complex morphology and is difficult to clean. So, it is important to bring irrigants into contact with the entire canal surfaces along its total micro anatomic complexity for effective action especially in the apical portions .

Irrigating solutions used during endodontic handling act through direct contact with the targeted bacteria. However, irrigants have inadequate penetration depth. It is highly desirable that chemical substances selected as endodontic irrigants have antimicrobial and organic tissue dissolution properties besides serving in the debridement of the root canal system and not being toxic to the tissues .Sodium hypochlorite (NaOCl) has been the gold standard for irrigation because of its ability to dissolve organic matter and high antimicrobial potential.

Conventional needle irrigation is the most commonly employed technique for delivering irrigants into the root canal system. However, the disadvantage of conventional needle irrigation is its passive action, and inability to deliver solutions into the narrow anatomical features of the root canal system. Despite the high success rates of root canal treatment, reducing the bacterial load below the level that is required to assure healing has become the accepted goal. Hence, several irrigant activation systems have been developed to increase the effectiveness of irrigation by providing energy within the canal to disperse and move the irrigant around the canal system in anticipation of them removing biofilm more effectively.

Therefore, various activation and agitation systems have been introduced to improve the irrigation penetration and effectiveness. These systems include manual dynamic agitation, sonic, passive ultrasonic, photon initiated photoacoustic streaming (PIPS), laser, XP-endo Finisher file, and Easy-Clean (EC).

The XP-endo Finisher file is a new rotary file presented to be used after root canal instrumentation as a final step in order to improve irrigant penetration and root canal cleaning and disinfection. It is made from a special nickel-titanium (NiTi) MaxWire alloy Hence, it possesses the shape memory effect when inserted into the canal (M-phase changed to A-phase) and exhibits superelasticity during canal preparation.

EC is an irrigation activating device, using an acrylonitrile butadiene styrene plastic instrument designed to produce vigorous intracanal fluid agitation.It has advantages of promoting agitation along the whole length of the instrument with no risk of deforming the canal walls.

There are many methods to evaluate penetration of irrigant solution into root canal but most them laboratory or ex-vivo using dye marker as Rhodamine B stain and methylene blue, while other radiopaque marker as Iohexol are used clinically.

Radiopaque contrast media as Iohexol can be used to assess the effect of various irrigation activating techniques on irrigant penetration into root canals in vivo as they can be seen in dental radiographs. Iohexol has the advantage of being a low osmolality agent that it is readily available in a sterile, pyrogen-free, nontoxic solution. It is widely used for angiocardiographic studies, thoracic and lumbar myelography, and in contrast enhancement for brain computed tomography and imaging of salivary glands.

Activation of irrigantion was considered one important method of bacterial reduction beside decreasing biofilm formation in root canals. on the other hand, it was reported that the activation protocols facilitate the disinfection of anatomical complexities and dentinal tubules.

According to the current knowledge, there is few studies concerning the effect of different irrigation activation techniques on enhancing irrigant penetration into the apical third of root canals and on reducing microbial infection, so this study aims to evaluate irrigant penetration depth and microbial reduction after using different irrigation activation techniques.

ELIGIBILITY:
Inclusion Criteria:

* • Asymptomatic vital/non vital teeth requiring root canal treatment.

  * Teeth with sound periodontal apparatus.
  * Teeth without pus or inflammatory exudates draining through the canal.
  * Teeth without anatomic variations.
  * Teeth with sinus tract.

Exclusion Criteria:

* • Patients with any systemic diseases.

  * Pregnant or lactating patients.
  * Immunocompromised patients.
  * Apparently thin roots in which apical preparation with #40 or #50 file would be overzealous.
  * Patient allergic to anything used in this procedure especially rubber dam material and Iohexol (radiographic contrast media).

Retreatment cases. Teeth with calcified canals.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
measurment of penetration depth of irrigant | at the same 1 day visit
  measurment the difference between the working length and penetration depth of irrigant
measurment of bacterial reduction following different irrigation activating techniques | 24-28 hours after culturing
  collection of 3 samples followed by culturing on blood agar and counting to calculate percentage of bacterial reduction

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mahmoud Farag, Phd, Principal Investigator — Professor of Endodontics; Dalia Abd Elhameed Sherif, Phd, Study Director — Lecturer of Endodontics; Kareman Ahmed Ebrahim Eshra, Phd, Principal Investigator — Professor of clinical Microbiology and Immunology
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreani Y, Gad BT, Cocks TC, Harrison J, Keresztes ME, Pomfret JK, Rees EB, Ma D, Baloun BL, Rahimi M. Comparison of irrigant activation devices and conventional needle irrigation on smear layer and debris removal in curved canals. (Smear layer removal from irrigant activation using SEM). Aust Endod J. 2021 Aug;47(2):143-149. doi: 10.1111/aej.12482. Epub 2021 Mar 8. PMID 33682268
- [Background] de Souza DS, S Silva AS, Ormiga F, Lopes RT, Gusman H. The effectiveness of passive ultrasonic irrigation and the easy-clean instrument for removing remnants of filling material. J Conserv Dent. 2021 Jan-Feb;24(1):57-62. doi: 10.4103/JCD.JCD_590_20. Epub 2021 Jul 5. PMID 34475681